CLINICAL TRIAL: NCT06518876
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Preliminary Efficacy, and Pharmacokinetic Characterization of KQ-2003 for Patients With Relapsed/Refractory POEMS Syndrome
Brief Title: A Study of KQ-2003 CAR-T Cell Therapy for Patients With Relapsed or Refractory POEMS Syndrome
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novatim Immune Therapeutics (Zhejiang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KQ-2003-BC101
Record Dates: First submitted 2024-07-08; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: POEMS Syndrome
MeSH Terms: conditions — POEMS Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase 1a: Low dose group (Experimental): Infusion of KQ-2003 CAR T-cells by single dose of 0.5×10^6 CAR-T cells/kg
  Interventions: Biological: KQ-2003 CAR T-cells
- Phase 1a: Medium dose group (Experimental): Infusion of KQ-2003 CAR T-cells by single dose of 1.0×10^6 CAR-T cells/kg
  Interventions: Biological: KQ-2003 CAR T-cells
- Phase 1a: High dose group (Experimental): Infusion of KQ-2003 CAR T-cells by single dose of 2.0×10^6 CAR-T cells/kg
  Interventions: Biological: KQ-2003 CAR T-cells
- Phase 1b: RP2D (Experimental): After all subjects in the Phase 1a dose-escalation study completed DLT observation, RP2D was determined based on the analysis results for the phase 1b expansion study.
  Interventions: Biological: KQ-2003 CAR T-cells

INTERVENTIONS:
Biological: KQ-2003 CAR T-cells — KQ-2003 CAR T-cell therapy involves autologous chimeric antigen receptor T-cells, capable of targeting both human B cell maturation antigen (anti-BCMA CAR) and CD19 antigen molecules (anti-CD19 CAR) simultaneously as a cellular therapy.

SUMMARY:
This is a multicenter, open-label, dose-escalation/expansion phase 1 study to evaluate the safety, tolerability, pharmacokinetic/pharmacodynamic characteristics and determine the recommended dose of KQ-2003 CAR T-cells for patients with Relapsed/Refractory POEMS Syndrome

DETAILED DESCRIPTION:
The study included the phase 1a dose escalation study and the phase 1b cohort extension study. The phase 1a study is an open, dose-escalation design with 3 dose groups according to the "3+3" dose escalation rule: low dose group (0.5×10^6 CAR T cells/kg), medium dose group (1.0×10^6 CAR T cells/kg), high dose group (2.0×10^6 CAR T cells/kg). After initial confirmation of maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D), a phase 1b cohort extension study will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old, male or female;
* Diagnosis of POEMS syndrome with relapsed or refractory disease;
* Eastern Cooperative Oncology Group (ECOG) Performance ≤2 ;
* Adequate venous access for the apheresis of peripheral blood mononuclear cell;
* Vascular Endothelial Growth Factor (VEGF) ≥1200ng/L；
* Overall Neuropathy Limitations Scale (ONLS) ≥ 1;
* Adequate organ function;
* Able and willing to comply with the study protocol and follow-up plan, and sign the informed consent form in writing.

Exclusion Criteria:

* Subjects who had previously received BCMA-CD19 dual-target CAR-T cell products or autologous stem cell transplantation within 12 weeks before the collection of peripheral blood mononuclear cells;
* Known allergy or hypersensitivity reactions to cyclophosphamide, fludarabine, dimethyl sulfoxide (DMSO), CD19, or BCMA-targeted drugs;
* Received any treatment that might influence the activity of CAR-T cells prior to the collection of peripheral blood mononuclear cells;
* Have history of vaccination within the 4 weeks preceding the collection of peripheral blood mononuclear cells;
* Have tested positive for cytomegalovirus and/or mycobacterium tuberculosis, or had any uncontrolled active infection within 14 days prior to the collection of peripheral blood mononuclear cells;
* Subjects infected with active HBV or HCV, HIV, syphilis;
* Subjects with known central nervous system disease, for example, seizure disorders, clinically significant cerebral ischemia/hemorrhage, dementia);
* Subjects currently experiencing active autoimmune diseases; Diagnosed with immunodeficiency or receiving any other form of immunosuppressive therapy within 7 days prior to enrollment in this study;
* Subjects with active bleeding or VTE events (such as pulmonary embolism or deep vein thrombosis) require anticoagulation;
* Have following severe diseases: unstable angina, cerebrovascular accident or transient ischemic attack, myocardial infarction , New York Heart Association (NYHA) Class ≥ III, congestive heart failure, poorly controlled severe arrhythmias or other cardiac diseases requiring mechanical support; subjects with known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal; subjects with known moderate or severe persistent asthma, or a history of asthma within the past 2 years, or currently having any category of uncontrolled asthma; subjects requiring oxygen to maintain adequate oxygen saturation; subjects with hypertension whose blood pressure cannot be lowered to the following range despite treatment with two or more antihypertensive medications;
* Have active malignancies;
* Have any non-hematologic toxicity resulting from prior treatments that cannot be restored to ≤ grade 1 or baseline, excluding alopecia and grade 2 neuropathy;
* Subjects had participated in other clinical trials and used its investigational drugs within the 3 months prior to the collection of peripheral blood mononuclear cells;
* History of alcohol abuse, drug addiction, substance abuse, or mental illness within the past year;
* Pregnant or lactating women;
* Any situation that the investigator believes may increase the risk of subjects or interfere with the results of clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-08-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with dose-limiting toxicity (DLT) | Within 28 days of receiving KQ-2003 CAR T-cells transfusion therapy
  For DLT evaluation, severity (grade) is classified according to common terminology criteria for adverse events version 5.0 (CTCAE v5.0).
Adverse Event | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  Safety will be assessed by adverse events (AEs), which include clinically significant abnormalities identified during a medical test (e.g. laboratory tests, electrocardiogram, vital signs, physical examinations). AEs will be coded by Medical Dictionary for Regulatory Activities (MedDRA) and their severity will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE, version 5.0).
Maximum Tolerated Dose (MTD) | Within 28 days of receiving KQ-2003 CAR T-cells transfusion therapy
  At least 6 subjects in the MTD dose group must complete the DLT assessment.
Recommended Phase 2 Dose (RP2D) | Through study completion, an average of 1 year
  To determine after all subjects in the Phase 1 dose-escalation study completed DLT observation

SECONDARY OUTCOMES:
Response of serum vascular endothelial growth factor level(VEGF) | Through study completion, an average of 2 years
  The improvements of serum VEGF will be assessed every three months by evaluating changes from baseline and will be described descriptively.
Hematologic response | Through study completion, an average of 2 years
  Hematologic response is also a criterion for assessing the efficacy of treatment for POEMS syndrome. The improvements of serum protein electrophoresis (SPEP) and immunofixation electrophoresis (IFE) will be assessed every three months by evaluating changes from baseline and will be described descriptively.
Response of positron emission tomography-scan (PET-CT) | Through study completion, an average of 2 years
  Observe the change in FDG uptake in the lesions of the subjects compared to the baseline, assessed every three months.
Response rate of critical organs | Through study completion, an average of 2 years
  Evaluate the changes in clinical symptoms compared to the baseline according to CTCAE 5.0. The assessment of clinical efficacy is conducted every three months after KQ-2003 CAR T-cells transfusion therapy.
Complete response rate (CRR) | Through study completion, an average of 2 years
  The definition of CRR is the proportion of subjects achieving CR confirmed by efficacy re-assessment after a minimum interval of three months.
Disease-free survival (DFS) | Through study completion, an average of 2 years
  DFS refers to time from treatment until the recurrence of disease (or death) after undergoing the study treatment.
Overall survival (OS) | Through study completion, an average of 2 years
  OS is the time from the start of cell infusion to the death of the subject.
Maximum concentration (Cmax) | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  Blood and bone marrow samples will be collected and used for pharmacokinetics assessments.
Time to maximum plasma concentration (Tmax) | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  Blood and bone marrow samples will be collected and used for pharmacokinetics
Levels of IL-2 | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  Blood samples will be collected and used for pharmacodynamic to evaluate the levels about cytokine levels
Levels of IL-6 | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  Blood samples will be collected and used for pharmacodynamic to evaluate the levels about cytokine levels
Levels of IL-10 | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  Blood samples will be collected and used for pharmacodynamic to evaluate the levels about cytokine levels
Levels of TNF-α | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  Blood samples will be collected and used for pharmacodynamic to evaluate the levels about cytokine levels
Levels of IFN-γ | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  Blood samples will be collected and used for pharmacodynamic to evaluate the levels about cytokine levels
Levels of C-reactive protein (CRP) | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  Blood samples will be collected and used for pharmacodynamic to evaluate the levels
Levels of ferritin | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  Blood samples will be collected and used for pharmacodynamic to evaluate the levels
CD19+B lymphocyte count | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  Blood samples will be collected and used for pharmacodynamic to evaluate the levels about peripheral blood lymphocyte subsets
CD20+B lymphocyte count | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  Blood samples will be collected and used for pharmacodynamic to evaluate the levels about peripheral blood lymphocyte subsets
CD3+T lymphocyte count | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  Blood samples will be collected and used for pharmacodynamic to evaluate the levels about peripheral blood lymphocyte subsets
CD4+T lymphocyte count | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  Blood samples will be collected and used for pharmacodynamic to evaluate the levels about peripheral blood lymphocyte subsets
CD8+T lymphocyte count | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  Blood samples will be collected and used for pharmacodynamic to evaluate the levels about peripheral blood lymphocyte subsets
ADA | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  The trial will evaluate the positive rate, titer and duration or persistence of ADA following the administration of CAR T-Cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences & Peking Union Medical College Hospital, Beijing, China